CLINICAL TRIAL: NCT00099918
Title: Efficacy and Safety of Vildagliptin Compared to Rosiglitazone in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2327
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to rosiglitazone in lowering overall blood glucose levels in people with type 2 diabetes who have not previously been treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* Not currently on drug therapy for type 2 diabetes
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular conditions
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2004-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 24 weeks
Adverse event profile after 24 weeks of treatment
Patients with endpoint HbA1c <7% at 24 weeks
Patients with reduction in HbA1c >/= 0.7% after 24 weeks
Change from baseline in HbA1c at 24 weeks for patients with high baseline HbA1c vs. low baseline HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Novartis Investigative Sites, Investigative Centers, Germany

REFERENCES:
- [Derived] Pratley RE, Schweizer A, Rosenstock J, Foley JE, Banerji MA, Pi-Sunyer FX, Mills D, Dejager S. Robust improvements in fasting and prandial measures of beta-cell function with vildagliptin in drug-naive patients: analysis of pooled vildagliptin monotherapy database. Diabetes Obes Metab. 2008 Sep;10(10):931-8. doi: 10.1111/j.1463-1326.2007.00835.x. Epub 2007 Dec 17. PMID 18093207
- [Derived] Pratley RE, Rosenstock J, Pi-Sunyer FX, Banerji MA, Schweizer A, Couturier A, Dejager S. Management of type 2 diabetes in treatment-naive elderly patients: benefits and risks of vildagliptin monotherapy. Diabetes Care. 2007 Dec;30(12):3017-22. doi: 10.2337/dc07-1188. Epub 2007 Sep 18. PMID 17878242
- [Derived] Rosenstock J, Baron MA, Dejager S, Mills D, Schweizer A. Comparison of vildagliptin and rosiglitazone monotherapy in patients with type 2 diabetes: a 24-week, double-blind, randomized trial. Diabetes Care. 2007 Feb;30(2):217-23. doi: 10.2337/dc06-1815. PMID 17259484